CLINICAL TRIAL: NCT01138696
Title: Long Term Follow-up of the "Stryker Dacron and Trevira Ligament" for ACL Repair
Brief Title: Long Term Follow-up of the "Stryker Dacron and Trevira Ligament" for Anterior Cruciate Ligament (ACL) Repair
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/670
Record Dates: First submitted 2010-04-22; First posted 2010-06-07 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: ACL Rupture; Replacement
Keywords: ACL
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stryker Dacron synthetic graft
  Interventions: Other: Questionnaires; Other: RX
- Trevira synthetic graft
  Interventions: Other: Questionnaires; Other: RX

INTERVENTIONS:
Other: Questionnaires — KOOS, IKDC, SF-36, Lysholm, Tegner, VAS),
Other: RX — X-rays and clinical investigation of the knee 20 years after surgery

SUMMARY:
About 20 years ago synthetic ligaments were used in orthopaedics / traumatology for the repairing and replacement of injuries of the anterior cruciate ligament. After less than 10 years it appeared that a relatively important number of patients showed complications on the basis of synovitis. The situation of another group of patients on the other hand evolved favourably without complications. The study to focuses on this group of patients and attempts to determine how the replacement without problems ab initio, evolved in the time.

It concerns a group of 57 patients who received an implantation in the UZ Ghent between November 85 and October 87 with the Stryker Dacron ligament and a group of 33 patients who received the Trevira ligament in the ASZ Aalst. The clinical result will be stipulated by means of standardized questionnaires and a clinical examination. The radiological result will be determined by the degree of integrity of the ligament that was implanted at the time. In this way the study could give an idea about the degree in which the technical success of the intervention correlates with the clinical success 20 years later.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received a Stryker Dacron or Trevira ligament to replace there ACL.
* Max age: 75
* Min age: 49
* Minimum follow up: 22 years

Ages: 49 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that received a Stryker Dacron or Trevira ligament to replace there ACL.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
to determine the evolution in pain, safety and tolerability of replacement of anterior cruciate ligament (ACL) after trauma or injury | 20 years after surgery
  Pain is measured by the VAS-score. For the evaluation of safety and tolerability the patients fill in the Tegner, Lysholm, IKDC, KOOS and SF-36 questionnaires

SECONDARY OUTCOMES:
A clinical and radiographical evaluation of the knee after implantation of a synthetic ligament. | 20 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: René Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be